CLINICAL TRIAL: NCT02676011
Title: Prevention of Brad Arrhythmia Induced by Repeated Succinylcholine by Atropine Sulfate During Gynecological Laparoscopic Surgery: a Randomized Controlled Trial
Brief Title: Brad Arrhythmia Induced by Repeated Succinylcholine During Gynecological Laparoscopic Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sayed Kaoud Abd-Elshafy, Associate Professor (Anesthesiology and Critical Care)- College of Medicine-Assiut University, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRB000087133
Record Dates: First submitted 2016-02-03; First posted 2016-02-05 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Bradycardia
Keywords: Atropine; Succinycholine; Laparoscopy; Gynecology
MeSH Terms: conditions — Bradycardia | interventions — Atropine; Succinylcholine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group A (Active Comparator): Intramuscular (IM) atropine (0.01 mg/kg) (1 ml) 30 minutes before induction of anesthesia, IV normal saline 10 ml 3 minutes before induction of anesthesia and normal saline mixed with second dose succinylcholine (1mg/kg) in 5 ml syringe with normal saline
  Interventions: Drug: IM atropine; Drug: IV normal saline; Drug: Normal saline mixed with second dose succinylcholine
- Group B (Active Comparator): 1 ml normal saline IM 30 minutes before induction of anesthesia, intravenously (IV) atropine (0.01 mg/kg) in 10 ml 3 minutes before induction of anesthesia and normal saline mixed with second dose succinylcholine (1mg/kg) in 5 ml syringe with normal saline
  Interventions: Drug: IV atropine; Drug: IM normal saline; Drug: Normal saline mixed with second dose succinylcholine
- Group C (Active Comparator): IM normal saline 1 ml normal 30 minutes before induction of anesthesia, IV normal saline 10 ml 3 minutes before induction of anesthesia and 1mg/kg atropine mixed with second dose succinylcholine (1mg/kg) in 5 ml syringe with normal saline
  Interventions: Drug: Atropine mixed with second dose succinylcholine; Drug: IM normal saline; Drug: IV normal saline
- Group D (Placebo Comparator): IM normal saline 1 ml normal 30 minutes before induction of anesthesia, IV normal saline 10 ml 3 minutes before induction of anesthesia and normal saline mixed with second dose succinylcholine (1mg/kg) in 5 ml syringe with normal saline
  Interventions: Drug: IM normal saline; Drug: IV normal saline; Drug: Normal saline mixed with second dose succinylcholine

INTERVENTIONS:
Drug: IM atropine — Atropine (0.01 mg/kg) (1 ml) IM 30 minutes before induction of anesthesia
  Other Names: IM atropine sulphate
  Arms: Group A
Drug: IV atropine — Atropine (0.01 mg/kg) intravenously (10 ml) 3 minutes before induction of anesthesia
  Other Names: IV atropine sulphate
  Arms: Group B
Drug: Atropine mixed with second dose succinylcholine — Atropine (0.01 mg/kg) added to the second dose succinylcholine (1mg/kg) prepared to 5 ml syringe with normal saline
  Other Names: atropine sulphate with succinylcholine
  Arms: Group C
Drug: IM normal saline — 1 ml normal saline IM 30 minutes before induction of anesthesia
  Other Names: Normal saline
  Arms: Group B; Group C; Group D
Drug: IV normal saline — IV 10 ml normal saline 3 minutes before induction of anesthesia
  Other Names: Normal saline
  Arms: Group A; Group C; Group D
Drug: Normal saline mixed with second dose succinylcholine — Second dose succinylcholine (1 mg/kg) prepared to 5 ml syringe with normal saline
  Other Names: Normal saline with succinylcholine
  Arms: Group A; Group B; Group D

SUMMARY:
Cardiac arrhythmias are a well-recognized complication of anesthesia for laparoscopy. The aim of this study was to evaluate the efficacy of atropine sulfate for prevention of brad arrhythmia induced by repeated succinylcholine during gynecological laparoscopic surgery.

DETAILED DESCRIPTION:
120 candidates, ASA 1 in the age range 18-40 years scheduled for elective diagnostic gynecological laparoscopic surgery were randomly assigned into 4 groups to receive either atropine sulfate or normal saline solution (as placebo).

ELIGIBILITY:
Inclusion Criteria:

* Female patients 18-50 years scheduled for elective diagnostic gynecological laparoscopic surgery

Exclusion Criteria:

* Cardiac
* Diabetes Mellitus
* Thyroid disease
* Any endocrine disease

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2016-02; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Occurrence of bradycardia | within the first 2 hours during surgery
  heart rate less than 60 per minutes or decrease more than 30% of baseline reading

SECONDARY OUTCOMES:
Nasopharyngeal secretion | within the first 4 hours during surgery
  suction of Nasopharyngeal secretion (ml) during and after extubation

CONTACTS AND LOCATIONS:
Overall Officials: sayed abd elshafy, M, Principal Investigator — associate professor
Locations (1):
- Faculty of Medicine, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided